CLINICAL TRIAL: NCT01719393
Title: Pulse Spectrum Analysis in Adult Asthmatics: Correlation With Lung Function, Asthma Control Exhaled Nitric Oxide and Metabolites in Exhaled Breath
Brief Title: Pulse Spectrum Analysis in Adult Asthmatics: Correlation With Lung Function, Asthma Control Exhaled Nitric Oxide and Metabolites in Exhaled Breath Condensate
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor-Investigator, National Taiwan University Hospital, M.D., National Taiwan University Hospital
Other Study IDs: 201207062RIC
Record Dates: First submitted 2012-10-30; First posted 2012-11-01 (Estimated); Last update posted 2012-11-01 (Estimated); Status verified 2012-10

CONDITIONS: Pulse Spectrum Analysis; Pulmonary Function; FeNO; Metabolites
Keywords: Asthma; Pulse spectrum analysis; lung function; exhaled nitric oxide; metabolites; exhaled breath condensate
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Exhaled brath condensate
Oversight: Data Monitoring Committee: No

SUMMARY:
Our hypothesis is that radial arterial pulse may reflect the severity and airway function in asthmatics. The aims of this study are to investigate the pulse spectrim of the radial artery in adult asthmatics, and evaluate its correlation with airy inflammation an lung funtion in asthmatics.

DETAILED DESCRIPTION:
The microcirculation is directly involved in the cellular matabolism and homeostasis. Our hypothesis is that radial arterial pulse spectrum may reflect the airway condition in asthmatics. The aims of this study are to investigate the pulse spectrim of the radial artery in adult asthmatics, and evaluate its correlation with lung function, asthma control status,exhaled nitric oxide, and metabolites in the exhaed breath condensates.

ELIGIBILITY:
Inclusion Criteria:

* Meet the diagnostic criteria of GINA guideline asthma patients

Exclusion Criteria:

* Cancer or immune impaired patients;
* pack-year smoking> 5;
* long-term ventilator-dependent patients
* Control group: 30 age matched healthy controls

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Asthma paitients
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2012-11; Primary Completion 2013-11 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Pulse spectral analysis | one year

CONTACTS AND LOCATIONS:
Overall Officials: Ping-Hung Kuo, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan